CLINICAL TRIAL: NCT04632459
Title: Phase II Study of Pembrolizumab Plus Ramucirumab in Metastatic Gastric or GEJ Adenocarcinoma as Salvage Treatment
Brief Title: Pembrolizumab Plus Ramucirumab in Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-03-115
Record Dates: First submitted 2020-09-04; First posted 2020-11-17 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab; Ramucirumab

STUDY DESIGN:
Intervention Model Description: Pembrolizumab Plus Ramucirumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pembrolizumab plus ramucirumab (Experimental): * Ramucirumab 8mg/kg on q2W
  * Pembrolizumab 200mg on q3W (pembrolizumab first followed by ramucirumab when concurrently administered on the same day)
  * If ramucirumab had to be stopped due to intolerable toxicity, pembrolizumab will be continued until unacceptable toxicity, disease progression or upto 35 cycles
  Interventions: Drug: pembrolizumab plus ramucirumab

INTERVENTIONS:
Drug: pembrolizumab plus ramucirumab — Patients will continue to receive study treatment, until they demonstrate objective disease progression (determined by modified RECIST 1.1) or until they meet any other discontinuation criteria.
  * Ramucirumab 8mg/kg on q2W
  * Pembrolizumab 200mg on q3W (pembrolizumab first followed by ramucirumab when concurrently administered on the same day)
  * If ramucirumab had to be stopped due to intolerable toxicity, pembrolizumab will be continued until unacceptable toxicity, disease progression or upto 35 cycles.

SUMMARY:
1. Objective 1) Primary Objective: To estimate preliminary overall response rate (ORR) of combination therapy of Ramucirumab and Pembrolizumab in patients with metastatic gastric or GEJ adenocarcinoma 2)Secondary Objectives: To assess secondary measures of clinical efficacy

   * Best Overall Response Rate: BORR
   * Disease Control Rate: DCR
   * Progression-Free Survival:PFS
   * Overall Survival: OS
   * Duration of Overall Response: DOR & maximal tumor shrinkage
2. Subjects : Patients with metastatic gastric or GEJ adenocarcinoma
3. Study design(Dosage & Treatment) Patients will continue to receive study treatment, until they demonstrate objective disease progression (determined by modified RECIST 1.1) or until they meet any other discontinuation criteria.

   * Ramucirumab 8mg/kg on q2W
   * Pembrolizumab 200mg on q3W (pembrolizumab first followed by ramucirumab when concurrently administered on the same day)
   * If ramucirumab had to be stopped due to intolerable toxicity, pembrolizumab will be continued until unacceptable toxicity, disease progression or upto 35 cycles.

DETAILED DESCRIPTION:
Goal : To estimate efficacy and safety of combination therapy of Ramucirumab and Pembrolizumab in patients with metastatic gastric or GEJ adenocarcinoma

Planned Sample Size : A maximum of 35 patients will be recruited to this single-arm phase II trial. In this single-arm phase II trial, 33 people were calculated using Simon's two-stage design and a total of 35 patients will be recruited to account for a 5% dropout rate.

The sample size is calculated by use of a two-stage minimax Simon's design to control the type I error at 2.5 % for null hypothesis that, for arm, the true response was 15 % or below and to have 90 % of power if the true response was 40 % or higher. 19 evaluable patients are to be treated in the first stage. If 3 or fewer response are observed in the first stage, the arm will be stopped. If at least 4 responses are observed in the first stage, 14 additional evaluable patients are to be entered onto the second stage. At the final analysis, the null hypothesis will be rejected if at least 9 responses are observed in 33 evaluable patients. RR is reported with its exact 95% CI.

Durationof Study: About 2 years from approval from the regulatory authority

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥18 years of age.
* The patient who has received an adequate information and provided informed consent for all the study-specific procedures in advance
* The patient has histologically or cytologically confirmed gastric carcinoma, including gastric adenocarcinoma or GEJ adenocarcinoma. (Patients with adenocarcinoma of the distal esophagus are eligible if the primary tumor involves the GEJ.) patient has metastatic disease or locally recurrent, unresectable disease.
* The patient's tumor tissue must have the pre-defined characteristics as follows ; EBV+ or PDL1 CPS≥10
* The patient has measureable or evaluable disease as determined by standard computed tomography (CT) or magnetic resonance imaging (MRI) imaging. Examples of evaluable, nonmeasurable disease include gastric, peritoneal, or mesenteric thickening in areas of known disease, or peritoneal nodules that are too small to be considered measurable by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* The patient has experienced disease progression during first-line treatment or second-line therapy for metastatic disease

  * Acceptable prior chemotherapy regimens for this protocol are combination chemotherapy regimens that include platinum and/or fluoropyrimidine components (acceptable prior platinum agents are cisplatin, carboplatin, or oxaliplatin; acceptable prior fluoropyrimidine agents are 5-FU, capecitabine, or S-1). Regimens including a third agent, such as an anthracycline or a taxane, are acceptable provided a fluoropyrimidine and/or a platinum were used.
  * Recurrence during or within 6 months of completion of adjuvant chemotherapy (capecitabine, 5-FU, or TS-1) will be considered as first-line chemotherapy.
* No prior exposure to anti-PD1 antibody or ramucirumab
* the patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
* Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

Hemoglobin ≥9.0 g/dL Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥100 x 109/L Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) AST (SGOT)/ALT (SGPT) ≤ 3.0 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN Serum creatinine ≤1.5 x institutional ULN urinary protein is ≤1+ on dipstick or routine urinalysis (INR) ≤1.5 and (PTT) ≤5 seconds above the ULN (unless receiving anticoagulation therapy). Patients on anticoagulation therapy with unresected primary tumors or local tumor recurrence following resection are not eligible

* Female patients of childbearing potential must have a negative pregnancy test (urine or serum), must not be breastfeeding and using adequate contraceptive measures.

Female patients must use a highly effective contraceptive measure from screening until 90 days after the last dose of drug. All methods of contraception (except for total abstinence) should be used in combination with the use of a condom by a male sexual partner for intercourse (see Restrictions below). (or vasectomy)

Female patients must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

1. Post-menopausal women defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatment.
2. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.

   1. . For the duration of the study and for 1 week after the last study drug administration, sexually active male patients must be willing to use barrier contraception i.e. condoms with all sexual partners. Where the sexual partner is a 'women of child-bearing potential' who is not using effective contraception, men must use a condom (with spermicide) during the study and for 6 months after the last dose of a study drug. (or vasectomy)

      -Biopsy during the screening window prior to dosing and at progression (if clinically feasible)

      Exclusion Criteria:

      -The patient has documented and/or symptomatic encephalitis, brain or leptomeningeal metastases.

      -The patient has experienced any Grade 3 to 4 GI bleeding within 3 months prior to enrollment.

      -The patient has experienced myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to enrollment.

      -The patient has a history of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy.

      -The patient has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the treating physician.

      -The patient has ongoing or active psychiatric illness or social situation that would limit compliance with treatment

      -The patient has uncontrolled or poorly controlled hypertension (>160 mmHg systolic or >100 mmHg diastolic for >4 weeks) despite standard medical management.

      -The patient has a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment.

      -The patient has received chemotherapy, radiotherapy, immunotherapy, or targeted therapy for gastric cancer within 2 weeks prior to enrollment.

      -The patient has received any investigational therapy within 30 days prior to enrollment.

      -The patient has undergone major surgery within 28 days prior to enrollment, or subcutaneous venous access device placement within 7 days prior to enrollment.

      -The patient has received prior therapy with an agent that directly inhibits VEGF (including bevacizumab), or VEGF Receptor 2 activity, or any antiangiogenic agent and immunotherapy.

      -The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti- inflammatory drugs (NSAIDs; including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.

      -The patient has a known allergy to any of the treatment components.

      -Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.

      -Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
      * Has an active infection requiring systemic therapy.
      * Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). 19. Has known active Hepatitis B or Hepatitis C (e.g., HCV RNA [qualitative] is detected) and liver cirrhosis. Chronic HBV infection with anti-viral agent prophylaxis is allowed.

        20. Has known liver cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.

        21. The patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24months
  Modified RECIST 1.1 criteria will be used to assess patient response to treatment by determining PFS and ORR. The modified RECIST 1.1 guidelines for measurable, non-measurable, target and non-target lesions and the objective tumour response criteria

SECONDARY OUTCOMES:
Best Overall Response Rate (ORR) | 24months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No